CLINICAL TRIAL: NCT06349525
Title: Retention of Telescopic Versus Locator Attachments And Marginal Bone Loss Surrounding Implants Supporting Maxillary Over-dentures: Two Year Randomized Clinical Trial
Brief Title: Retention of Telescopic Versus Locator Attachments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Delta University for Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DU-2021-00103
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-03

CONDITIONS: Jaw, Edentulous
Keywords: edentulous; Maxillary implant supported overdenture; Retention; Marginal bone loss; Locator; Telescopic
MeSH Terms: conditions — Jaw, Edentulous; Mouth, Edentulous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 implants overdenture with telescopic (Experimental): Completely edentulous maxillary arch treated with 4 implants overdenture
  Interventions: Device: telescopic overdenture
- 4 implant supported overdenture with Locator (Active Comparator): Completely edentulous maxillary arch treated with 4 implant supported overdenture
  Interventions: Device: Locator overdenture

INTERVENTIONS:
Device: telescopic overdenture — Maxillary implant supported telescopic overdenture
  Arms: 4 implants overdenture with telescopic
Device: Locator overdenture — Maxillary implant supported locator overdenture
  Arms: 4 implant supported overdenture with Locator

SUMMARY:
Forty patients ( 24female and16 male )with completely edentulous maxilla and mandible . All patients received implant supported mandibular and maxillary overdentures. The patients were randomly divided into two groups according to attachments retaining Max IOD that supported by four axial implants in maxilla . The TA was used to retain group I (GrI) MaxIOD , while that of group II (Gr II) was retained by LA. MaxIOD retention and MBL(vertical and horizontal) around implants of both groups was recorded at time of insertion (R0) ,then twelve(R12)and (R24) months following insertion of the prosthesis.

DETAILED DESCRIPTION:
Parallel groups, two arms, randomized controlled trial (RCT) with 1:1 allocation ratio was designed, retention of telescopic attachment and locator attachment among patients with completely edentulous maxillary arch and intended to use maxillary overdenture was compared. The minimum proper sample size was 20 participants in each group to be able to detect a real difference in retention equal to 2 N with 80% power at α = 0.05 level using Student's t test for independent samples.

The stone casts were poured and mounted guided by the the occlusion of upper and lower dentures in centric relation to evaluate inter-arch distance. Pre-operative panorama was initially made to assess bone quality and quantity of edentulous maxillary ridge New Complete maxillary and mandibular dentures were made using semi-anatomic teeth arranged following balanced occlusion . The stent is scanned in the patient's mouth using CBCT. DICOM (digital imaging and communications in medicine) was applied for the virtual planning of the implants using exocad software .

Two virtual implant models were used and their criteria are mentioned (in table 2). Implants were planned at lateral-canine areas equidistant from midline and another two implants at first molar bilaterally . A safety zone of a minimum of 2 mm between the implants and vital structures like the maxillary sinus was planned Surgical procedure Two stage surgical protocol was followed for insertion of implants for both groups in their planned position via the same oral and maxillofacial surgeon. Presurgical prophylactic medications were prescribed, including: 1gm Augmentin®, prednisone, and 0.2% chlorhexidine digluconate started 8 hours before surgery and continued for 7 days following surgery. Analgesic drug was prescribed once daily or when needed. Flapless surgical technique was followed guided by mucosa-supported surgical stents that were checked intraorally for stability and fitness. The stents were fixed to the bone using three fixation screws. Implants were inserted at a minimum of 35 Ncm torque. After complete insertion of fixtures and screwing of covering abutments , tissue conditioner was used for relining and fitting of the existing maxillary denture to the mucosa. Participants were instructed to eat a soft diet and perform oral hygiene procedures.

ELIGIBILITY:
Inclusion Criteria:

* have sufficient bone volume(classes IV to VI, Cawood and Howell) and quality (classes I to III, Lekholm and Zarb)
* be fully edentulous for at least 1 year and did not have an American Society of Anesthesiologists score (ASA) of IV or higher.
* be with Angle Class I maxillo- mandibular relationship
* have Adequate zone of keratinized attached mucosa >5mm over the crest of the upper and lower ridge
* have adequate inter-arch space (22 mm) as determined by the mounted casts carrying the patient upper and lower complete dentures .

Exclusion Criteria:

* Any medical disorders that could complicate the surgical phase or affect osseointegration as osteoporosis, uncontrolled diabetes and hypertension
* Smoking; - Former radiotherapy in the head and neck region
* Former pre-prosthetic surgery or loss of implants in the maxilla
* Patients with para-functional habits (as clenching or bruxism)
* Hard tissue augmentation / grafting.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Retention | 1 month, 12 months, and 24 months
  Retention was measured by a digital force gauge device (Extech's Model 475055 Digital Force Gauge FLIR Commercial Systems, Inc.) that measures tension or compression force (pull/push) to values of up to 980 Newton.25 The snap hook of the device engaged a screw fixed to the geometric center of denture bases using self-cure acrylic resin. Then pulling action was applied till the denture separation recording the amount of retention in Newton.

SECONDARY OUTCOMES:
Marginal bone loss | 12 months and 24 months
  Digital periapical radiographs were made using a direct digital imaging system (Digora Optime, Orion Corp./Soredex). Standardization of film position was done by fixing the film positioner to the implants using the placement aid of the implants. The digital images were traced using the accompanying software, and vertical and horizontal bone losses were measured

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa I Ibrahim, Principal Investigator — Assoc. Prof.
Locations (1):
- Delta University for Science & Technology, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No